CLINICAL TRIAL: NCT03206970
Title: A Single-Arm, Open-Label, Multicenter Phase 2 Study to Evaluate Efficacy and Safety of BGB-3111, a Bruton's Tyrosine Kinase (BTK) Inhibitor, in Subjects With Relapsed or Refractory Mantle Cell Lymphoma (MCL)
Brief Title: Study to Evaluate Efficacy and Safety of BGB-3111 in Participants With Relapsed or Refractory Mantle Cell Lymphoma (MCL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-206; CTR20160888 (Registry Identifier: Center for drug evaluation, CFDA)
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Results first posted 2020-05-13 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Refractory Mantle Cell Lymphoma; Relapsed Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib (Experimental): Zanubrutinib (160 milligrams) administered orally twice daily
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — Administered as specified in the treatment arm.
  Other Names: BGB-3111

SUMMARY:
The primary objective of this study was to evaluate the efficacy of zanubrutinib in participants with centrally confirmed relapsed or refractory MCL.

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnostic report had to include evidence for morphological and cyclin D1 or t (11; 14).
2. Eastern Cooperative Oncology Group performance status of 0-2.
3. Measurable disease by computed tomography/magnetic resonance imaging.
4. Received prior regimens for MCL.
5. Documented failure to achieve any response, (stable disease or progressive disease during treatment) or documented progressive disease after response to the most recent treatment regimen.
6. Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x upper limit of normal (ULN).
7. Total bilirubin ≤ 2 x ULN (unless documented Gilbert's syndrome).
8. Life expectancy of > 4 months.

Key Exclusion Criteria:

1. Current or history of central nervous system lymphoma.
2. Prior exposure to a BTK inhibitor before enrollment.
3. Prior corticosteroids with anti-neoplastic intent within 7 days.
4. Major surgery within 4 weeks of screening.
5. Toxicity must have recovered from prior chemotherapy.
6. History of other active malignancies within 2 years of study entry.
7. Currently clinically significant active cardiovascular disease.
8. QT interval corrected with Fridericia's formula > 450 microseconds or other significant electrocardiogram abnormalities.
9. Uncontrolled systemic infection or infection requiring parenteral anti-microbial therapy.
10. Known human immunodeficiency virus infection, or active hepatitis B or hepatitis C infection (detected positive by polymerase chain reaction).

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2020-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — BeiGene
Locations (13):
- China (13):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Institute of Hematology and Hospital of Blood Disease, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Yuqin Song, Keshu Zhou, Dehui Zou, Jianfeng Zhou, Jianda Hu, Haiyan Yang, Huilai Zhang, Jie Ji, Wei Xu, Jie Jin, Fangfang Lv, Ru Feng, Sujun Gao, Daobin Zhou, Haiyi Guo, Aihua Wang, James Hilger, Jane Huang, William Novotny, Muhtar Osman, Jun Zhu; Safety and Activity of the Investigational Bruton Tyrosine Kinase Inhibitor Zanubrutinib (BGB-3111) in Patients with Mantle Cell Lymphoma from a Phase 2 Trial. Blood 2018; 132 (Supplement 1): 148. doi: https://doi.org/10.1182/blood-2018-99-117956
- [Result] Song Y, Zhou K, Zou D, Zhou J, Hu J, Yang H, Zhang H, Ji J, Xu W, Jin J, Lv F, Feng R, Gao S, Guo H, Zhou L, Elstrom R, Huang J, Novotny W, Wei R, Zhu J. Treatment of Patients with Relapsed or Refractory Mantle-Cell Lymphoma with Zanubrutinib, a Selective Inhibitor of Bruton's Tyrosine Kinase. Clin Cancer Res. 2020 Aug 15;26(16):4216-4224. doi: 10.1158/1078-0432.CCR-19-3703. Epub 2020 May 27. PMID 32461234
- [Result] Tam CS, Opat S, Simpson D, Cull G, Munoz J, Phillips TJ, Kim WS, Rule S, Atwal SK, Wei R, Novotny W, Huang J, Wang M, Trotman J. Zanubrutinib for the treatment of relapsed or refractory mantle cell lymphoma. Blood Adv. 2021 Jun 22;5(12):2577-2585. doi: 10.1182/bloodadvances.2020004074. PMID 34152395
- [Derived] Moslehi JJ, Furman RR, Tam CS, Salem JE, Flowers CR, Cohen A, Zhang M, Zhang J, Chen L, Ma H, Brown JR. Cardiovascular events reported in patients with B-cell malignancies treated with zanubrutinib. Blood Adv. 2024 May 28;8(10):2478-2490. doi: 10.1182/bloodadvances.2023011641. PMID 38502198
- [Derived] Song Y, Zhou K, Zou D, Zhou J, Hu J, Yang H, Zhang H, Ji J, Xu W, Jin J, Lv F, Feng R, Gao S, Guo H, Zhou L, Huang J, Novotny W, Kim P, Yu Y, Wu B, Zhu J. Zanubrutinib in relapsed/refractory mantle cell lymphoma: long-term efficacy and safety results from a phase 2 study. Blood. 2022 May 26;139(21):3148-3158. doi: 10.1182/blood.2021014162. PMID 35303070

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 14 study centers in China; 13 study centers enrolled participants. Once the primary and secondary objectives were met and the analysis was complete, sponsor ended the study on 08 September 2020 and transferred all participants remaining on treatment to long term extension study.
Groups:
- Zanubrutinib: Zanubrutinib (160 milligrams [mg]) administered orally twice daily (BID) until disease progression, unacceptable toxicity or death, withdrawal of consent, lost to follow up, or study termination by sponsor, which comes first.
Period: Overall Study
Arm/Group | Zanubrutinib
Started | 86
Received at Least 1 Dose of Study Drug (Safety Analysis Set) | 86
Completed | 0
Not Completed | 86
Not completed — Death | 21
Not completed — Withdrawal by Subject | 13
Not completed — Lost to Follow-up | 3
Not completed — Primary and secondary objectives were met and remaining participants transferred to LTE by sponsor | 49

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All participants who received any dose of study drug.
Groups:
- Zanubrutinib: Zanubrutinib (160 mg) administered BID until Zanubrutinib (160 milligrams [mg]) administered orally twice daily (BID) until disease progression, unacceptable toxicity or death, withdrawal of consent, lost to follow up, or study termination by sponsor, which comes first.
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (8.18)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 64
  ≥ 65 years | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 86
Region of Enrollment [Number; unit: participants]
  China | 86
Mantle Cell Lymphoma (MCL) Disease Stage at Study Entry [Count of Participants; unit: Participants] — Participants' MCL disease stage at consent date, with higher stages indicating more severe MCL.
  Participants
    MCL Stage I | 1
    MCL Stage II | 7
    MCL Stage III | 14
    MCL Stage IV | 64
Disease Status [Count of Participants; unit: Participants]
  Relapsed Disease | 41
  Refractory Disease | 45
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — Grade 0 = Fully active, able to carry on all pre-disease performance without restriction; Grade 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg, light house work, office work; Grade 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; Lower grades indicate better outcome.
  Participants
    Grade 0 | 60
    Grade 1 | 22
    Grade 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) As Assessed By Independent Review Committee
Description: The ORR was assessed in accordance with the 2014 modification of the International Working Group on non-Hodgkin Lymphoma Criteria. The ORR was defined as the percentage of participants achieving a best overall response (BOR) of complete response (CR) or partial response (PR). The BOR was defined as the best response recorded from the start of zanubrutinib until data cut or start of new antineoplastic treatment. Participants with no post-baseline response assessment (due to any reason) were considered non-responders for BOR.
Time Frame: Up to 1 year and 11 months
Population: Safety Analysis Set: All participants who received any dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Zanubrutinib: Zanubrutinib (160 mg) administered BID until disease progression, unacceptable toxicity or death, withdrawal of consent, lost to follow up, or study termination by sponsor, which comes first.
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 86
Participants | 72
Statistical Analysis 1: Comparison: Zanubrutinib; A binomial exact test was performed to test against the null hypothesis H0: ORR=0.40 using the significant level of 0.025 (1-sided); Test type: Other; p < .0001, Binomial Exact Test; Clopper-Pearson = 83.7, 95% CI 2-sided [74.2 to 90.8]

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from the starting date of zanubrutinib to the date of first documentation of disease progression or death, whichever occurred first. Participants who did not have disease progression were censored at their last valid tumor assessment. A six-month progression-free survival rate was defined as no disease progression after treated with zanubrutinib for over six months (under control). The 95% confidence interval (CI) lower bound was 33.1 months while the upper bound could not be estimated.
Time Frame: Up to 3 years and 6 months
Population: Safety Analysis Set: All participants who received any dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 86
months | 33.0 [19.4 to NA] — NA = Not estimable due to insufficient number of participants with events

3. Secondary Outcome: Time To Response
Description: Time to response was defined as the time from treatment initiation to the first documentation of response.
Time Frame: Up to 3 years and 6 months
Population: Safety Analysis Set: All participants who received any dose of study drug.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 72
months | 2.72 (0.105)

4. Secondary Outcome: Duration Of Response
Description: The duration of response was defined as the time from the date that the response criteria are first met to the date that Progressive Disease was objectively documented or death (whichever occurs first). Participants who did not have disease progression were censored at their last valid assessment.
Time Frame: Up to 3 years and 6 months
Population: Safety Analysis Set: All participants who received any dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 86
months | NA [24.9 to NA] — NA = Not estimable due to insufficient number of participants with events

5. Secondary Outcome: ORR As Assessed By The Investigator
Description: The ORR was assessed in accordance with the 2014 modification of the International Working Group on non-Hodgkin Lymphoma Criteria. The ORR was defined as the percentage of participants achieving a BOR of CR or PR. The BOR was defined as the best response recorded from the start of zanubrutinib until data cut or start of new antineoplastic treatment. Participants with no post-baseline response assessment (due to any reason) were considered non-responders for BOR. For this outcome measure, only investigator-assessed data are analyzed and reported because of the high rate of concordance between the Independent Review Committee and investigator assessments for the primary outcome measure of ORR.
Time Frame: Up to 3 years and 6 months
Population: Safety Analysis Set: All participants who received any dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 86
Participants | 72
Statistical Analysis 1: Comparison: Zanubrutinib; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Binomial Exact Test; Clopper-Pearson = 83.7, 95% CI 2-sided [74.2 to 90.8]

6. Secondary Outcome: Number Of Participants Experiencing Treatment -Emergent Adverse Events (AEs)
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study drug, whether considered related to study drug or not. A summary of serious and all other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
  A treatment-emergent adverse event (TEAE) is defined as an AE that had an onset date or a worsening in severity from baseline (pretreatment) on or after the date of first dose of study drug up to 30 days following study drug discontinuation (Safety Follow-up visit) or initiation of new anticancer therapy, whichever comes first.
Time Frame: From the initiation of study drug until 30 days after the last dose (Up to 3 years and 6 months)
Population: Safety Analysis Set: All participants who received any dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 86
Participants | 83

7. Secondary Outcome: Number Of Participants Experiencing AEs Leading To Treatment Discontinuation
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study drug, whether considered related to the study drug or not. A summary of serious and all other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: From the initiation of study drug until 30 days after the last dose (Up to 3 years and 6 months)
Population: Safety Analysis Set: All participants who received any dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 86
Participants | 8

ADVERSE EVENTS:
Time Frame: Day 1 through 3 years and 6 months
Description: Safety Analysis Set
Groups:
- Zanubrutinib: Zanubrutinib (160 mg) administered BID for over 3 years.
Arm/Group | Zanubrutinib
All-Cause Mortality (participants affected / at risk) | 7/86
Serious Adverse Events (participants affected / at risk) | 25/86
Other Adverse Events (participants affected / at risk) | 82/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zanubrutinib (N=86)
Anaemia (Blood and lymphatic system disorders) | 1
Bone marrow necrosis (Blood and lymphatic system disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Death (General disorders) | 2
Bronchitis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 10
Pneumonia fungal (Infections and infestations) | 1
Pneumonia klebsiella (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Ureterolithiasis (Renal and urinary disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zanubrutinib (N=86)
Anaemia (Blood and lymphatic system disorders) | 14
Leukopenia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 14
Toothache (Gastrointestinal disorders) | 6
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Oedema peripheral (General disorders) | 4
Peripheral swelling (General disorders) | 3
Pyrexia (General disorders) | 7
Asymptomatic bacteriuria (Infections and infestations) | 4
Folliculitis (Infections and infestations) | 3
Otitis media (Infections and infestations) | 4
Pharyngitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 33
Urinary tract infection (Infections and infestations) | 10
Viral upper respiratory tract infection (Infections and infestations) | 5
Alanine aminotransferase increased (Investigations) | 16
Aspartate aminotransferase increased (Investigations) | 9
Blood bilirubin increased (Investigations) | 4
Blood creatinine increased (Investigations) | 8
Blood immunoglobulin G decreased (Investigations) | 4
Blood urine present (Investigations) | 11
Lymphocyte count decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 39
Platelet count decreased (Investigations) | 28
Weight decreased (Investigations) | 4
Weight increased (Investigations) | 7
White blood cell count decreased (Investigations) | 29
Hyperglycaemia (Metabolism and nutrition disorders) | 12
Hyperuricaemia (Metabolism and nutrition disorders) | 12
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Insomnia (Psychiatric disorders) | 5
Haematuria (Renal and urinary disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 31
Hypertension (Vascular disorders) | 13
Pneumonia (Infections and infestations) | 7
Nasopharyngitis (Infections and infestations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 3
Chest discomfort (General disorders) | 3
Headache (Nervous system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT03206970/Prot_001.pdf
  • Statistical Analysis Plan (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT03206970/SAP_000.pdf